CLINICAL TRIAL: NCT01063465
Title: Measurement of Mechanical Properties of the Healing Achilles Tendon With or Without Early Weightbearing in a Clinical Randomized Trial
Brief Title: Measurement of Mechanical Properties of the Healing Achilles Tendon With or Without Early Weightbearing
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Linkoeping University (Other Government)
Responsible Party: Thorsten Schepull, M.D., Orthopaedic department, University Hospital Linkoeping, Sweden
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 001
Record Dates: First submitted 2010-02-04; First posted 2010-02-05 (Estimated); Last update posted 2010-02-05 (Estimated); Status verified 2009-01

CONDITIONS: Achilles Tendon Rupture; Soft Tissue Injury; Tendon Injury
Keywords: Achilles; Tendon; weightbearing
MeSH Terms: conditions — Soft Tissue Injuries; Tendon Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early weightbearing (Experimental)
  Interventions: Device: Early weightbearing
- Control group (Experimental)
  Interventions: Device: Early weightbearing

INTERVENTIONS:
Device: Early weightbearing — Patients in the intervention group are after 2 weeks supposed to remove the cast twice a day and use a special training pedal for 5 weeks (until cast removal).

SUMMARY:
The purpose of this study is to measure the mechanical properties of healing Achilles tendons in humans after early controlled weightbearing, compared with a control group in a randomized, single-blinded trial. The mechanical properties are measured using radiostereophotogrammetic x-rays (RSA).

Hypothesis: Early weightbearing improves mechanical properties of the healing Achilles tendon.

DETAILED DESCRIPTION:
Patient with an acute Achilles tendon rupture coming to the local emergency room are asked to participate in our study. Patients have to be between 18 and 60 years and they must not have any contraindications for surgical treatment.

Patients who are interested in participating in the study receive oral and in written information about the study of the main investigator of the study (Thorsten Schepull). Patients who then agree to participate in the study are registered for surgery. All patients are operated the same way in local anaesthesia within 5 days after injury. We are going to use a conventional open technique with a dorso-medial approach. Tendon ends are going to be adapted with a resorbable suture and we are going to implant 2 Tantalum beads (size 0.8 mm) in the distal part of the tendon and 2 Tantalum beads with the same size in the proximal part. A short leg cast is going to be applied with the foot in the equinus position.

Randomization to early weightbearing or control group is done postoperatively

Group 1 (control group):

The short leg cast that is going to be applied during operation with the foot in the equinus position is removed after 3.5 weeks and a new cast is applied with the ankle in a neutral position for another 3.5 weeks. The new cast is removed after 3.5 weeks (cast treatment in total 7 weeks). Physiotherapy starts after cast removal, following our previous hospital routines. Full activity, including sports, is allowed after approximately 5 months.

We are going to perform RSA after 7 weeks (within 15 minutes after cast removal), after 19 weeks i.e. 12 weeks after cast removal, and after 52 weeks (12 months). A certain frame is used allowing us to apply a pedal to the forefoot and load it with weights. The first force applied to the pedal is 25 N and the second is 150 N. The same day CT scans of the injured Achilles tendon are taken.

Group 2 (early weightbearing):

The cast from surgery i removed after 2 weeks and replaced by a removable Air Cast Walker. The patient is provided with a special training pedal where pedal resistance can be increased during the treatment period. The patients are using the Air Cast Walker for 5 weeks (cast treatment in total 7 weeks), but is supposed to remove the cast twice a day and supposed to use the training pedal.

Follow-ups at 7 (cast removal), 19 and 52 weeks using RSA and CT are performed as in group 1.

ELIGIBILITY:
Inclusion Criteria:

* Acute Achilles Tendon rupture
* Age between 18 and 60 years

Exclusion Criteria:

* Previous rupture of either Achilles tendon
* Diabetes mellitus
* History of cancer
* History of Rheumatoid disease
* Treatment with steroids
* Any counterindication for surgical treatment

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35 (Estimated)
Dates: Start 2009-02; Primary Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Modulus of Elasticity | 7 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Linkoeping, Linköping, Sweden